CLINICAL TRIAL: NCT02024581
Title: A Multi-center, Double-blind, Placebo-controlled, Randomized Safety and Efficacy Trial of a Botanical Drug Product Containing East Indian Sandalwood Oil (EISO) for the Treatment of Molluscum Contagiosum in Pediatric Subjects
Brief Title: A Trial of a Botanical Drug Containing East Indian Sandalwood Oil (EISO) for the Treatment of Molluscum Contagiosum
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor chose to close
Sponsor: ViroXis Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIR003-01
Record Dates: First submitted 2013-12-19; First posted 2013-12-31 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Molluscum Contagiosum
Keywords: pediatric; dermatology; East Indian sandalwood oil; pox virus
MeSH Terms: conditions — Molluscum Contagiosum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10% East Indian sandalwood oil cream (Active Comparator): East Indian sandalwood oil in a cream formulation administered twice a day for ninety (90) days
  Interventions: Drug: 10% East Indian sandalwood oil cream
- Placebo cream (Placebo Comparator): A scented cream formulation administered twice a day for ninety (90) days
  Interventions: Drug: Placebo Cream

INTERVENTIONS:
Drug: 10% East Indian sandalwood oil cream — A topical oil/water emulsion cream containing 10% East Indian sandalwood oil (EISO)
  Other Names: Albuterpenoids; EISO
  Arms: 10% East Indian sandalwood oil cream
Drug: Placebo Cream — A sandalwood-scented oil/water emulsion topical cream matching the appearance of the active comparator creams
  Arms: Placebo cream

SUMMARY:
This trial will examine the safety, tolerability and efficacy of one strength of East Indian sandalwood oil (EISO) in a cream base compared to a placebo for treatment of molluscum contagiosum in pediatric subjects. Trial participants will be asked to apply study medication twice a day for sixty (60) days. Efficacy will be evaluated by clinical staff and patients will be asked to assess tolerability as well as any improvement experienced during the trial.

DETAILED DESCRIPTION:
This trial will be a multi-center, double-blind, randomized, placebo-controlled safety and efficacy trial to evaluate the efficacy and safety of VIR003 treatment regimen when administered to pediatric subjects with molluscum contagiosum.

Once subject eligibility is confirmed the subject will start the Treatment Period of the study. All subjects will receive active treatment or placebo with the first dose applied at the Day 0 Study Visit. Subjects will be instructed on how to apply the study medication twice a day for 90 days of treatment. Subjects will return to the clinic on Study Days, 7, 14, 30, 45, 60 and 90 for routine evaluations and then on Study Day 97 for the Final Study Visit.

Safety will be assessed by evaluating adverse events (AEs) with respect to severity, duration, and relationship to study drug. In addition tolerability evaluations will be performed at each study visit.

The preliminary efficacy evaluation for the study will be the resolution of molluscum contagiosum lesions at Study Day 90 in evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included in the trial if they meet all of the following criteria:

* Are between 2 and 17 years of age, inclusive, at screening.
* Have a diagnosis of molluscum contagiosum that is treatable with a topical agent and at least five (5) lesions on the treatment area.
* Are free of any systemic or dermatologic disorder, which, in the opinion of the investigator will interfere with the study results or increase the risk of adverse events.
* Are willing to refrain from using non-approved lotions, sunscreen, moisturizer, cleansers, cosmetics or creams on the affected areas during the treatment period.
* Whose parent or guardian is able to give written informed consent and potential pediatric subjects 7 years of age or older to provide assent in a manner approved by the Institutional Review Board and comply with the requirements of the study.

Exclusion Criteria:

Subjects will be excluded from the trial if they meet any of the following criteria:

* Are immunosuppressed.
* Have regular physical contact with a sibling or other person with molluscum contagiosum virus (MCV), unless that person is also enrolled in the study.
* Have used or are planning to use immunosuppressive or immunomodulatory medication (including oral or parenteral corticosteroids) in the previous 30 days.
* Are undergoing treatment or have been treated in the last 30 days prior to Screening with isotretinoin or any other type of topical therapy (e.g., corticosteroids, cantharidin, podophyllin, podofilox, iodine, salicylic acid, retinoids, diclofenac, hyaluronic acid, potassium hydroxide, imiquimod).
* Have used liquid nitrogen in the treatment area in the last 30 days prior to Screening.
* Have undergone curettage, electrocoagulation, taping or clamping of the infected area.
* Are taking antiviral medication including but not limited to cimetidine and cidofovir.
* Have any active skin malignancy or infection other than molluscum contagiosum.
* Have a molluscum contagiosum infection in an untreatable area (i.e., mucosal surfaces, anogenital, periorbital, and facial regions).
* Have any condition that in the opinion of the investigator would confound the safety and/or efficacy assessments.
* Have participated in any clinical trial in the previous 30 days.
* Have a known sensitivity to any of the constituents of the test product including sensitivities to sandalwood oil, fragrances or any member of the Compositae family of vascular plants (e.g., sunflowers, daisies, dahlias, etc.).
* Are pregnant, breastfeeding, or unwilling to practice an acceptable form of birth control during the study, if applicable.
* Have a present condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2016-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
Safety profile of the treatment | Monitored throughout the trial (90 Days)
  The primary purpose of this study is to determine the safety profile of VIR003. Safety will be assessed by evaluating adverse events (AEs) with respect to severity, duration, and relationship to study drug compared to placebo.

SECONDARY OUTCOMES:
Change in lesion count | Measured at Day 90
  Percent change in lesion count from Baseline to Study Day 90 in evaluable subjects
Improvement in GAIS score | Measured at Day 90
  Percentage of subjects who are very much improved, much improved, or improved (treatment success) at Day 90, as judged by the Global Aesthetic Improvement Scale (GAIS).
Complete resolution of lesions | Measured at Day 90
  1. The percentage of subjects with complete resolution of molluscum contagiosum lesion at Study Day 90 in evaluable subjects. The percentage of subjects with complete resolution of molluscum contagiosum lesion at Study Day 90 in evaluable subjects.
Improvement in Evaluator's Global Severity Score (EGSS) | Measured at Day 90
  Percentage of subjects with a baseline Evaluator's Global Severity Score (EGSS) of "moderate" or worse who are "clear" or "almost clear," or have at least a two-grade improvement at Day 90 as judged by the EGSS.

CONTACTS AND LOCATIONS:
Overall Officials: John C. Browning, MD FAAD FAAP, Principal Investigator — Texas Dermatology and Laser Specialists
Locations (1):
- Texas Dermatology and Laser Specialists, San Antonio, Texas, United States